CLINICAL TRIAL: NCT02725359
Title: Preemptive Single Dose Tizanidine and Ultrasound Guided Superficial Cervical Block on Pain After Thyroidectomy
Brief Title: Tizanidine and Superficial Cervical Block on Pain After Thyroidectomy
Acronym: PTUSGSCB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ali Ahiskalioglu, MD, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AUTF ANESTHESIA
Record Dates: First submitted 2016-03-21; First posted 2016-04-01 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Thyroidectomy
Keywords: Thyroidectomy pain; Tizanidine; Postoperative analgesia; Ultrasound guided Superficial cervical plexus block
MeSH Terms: interventions — tizanidine; Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Group Placebo (Group P) will receive placebo 1 hour before surgery and bilateral superficial cervical block with saline 10 ml each side
  Interventions: Drug: Placebo; Drug: Saline
- Tizanidine (Experimental): Group Tizanidine (Group T) will receive 6 mg tizanidine 1 hour before surgery and bilateral superficial cervical block with %0.25 bupivacaine 10ml each side
  Interventions: Drug: Tizanidine; Drug: Bupivacaine
- Bupivacaine (Active Comparator): Group Bupivacaine will receive placebo 1 hour before surgery and bilateral superficial cervical block with %0.25 bupivacaine 10ml each side
  Interventions: Drug: Placebo; Drug: Bupivacaine

INTERVENTIONS:
Drug: Placebo — Group Placebo: will receive a placebo pill 1 hour before surgery
  Other Names: Placebo pill
  Arms: Bupivacaine; Placebo
Drug: Tizanidine — Group T: 6 mg tizanidine1 hour before surgery
  Other Names: Sirdalud MR
  Arms: Tizanidine
Drug: Bupivacaine — Group Bupivacaine will receive USG guided SCPB with %0,25 bupivacaine bilaterally 10 ml each side
  Arms: Bupivacaine; Tizanidine
Drug: Saline — USG guided SCPB with saline bilaterally 10 ml each side
  Other Names: Saline block
  Arms: Placebo

SUMMARY:
Thyroid surgery is a quite painful procedure performed in a sensitive skin area of the human body. Unless pain is treated adequately thyroid surgery may cause severe postoperative pain and discomfort for the patients.

a2-Agonists are sympatholytic and centrally acting antihypertensive agents. In addition to their hypotensive effect, a2-agonists are also used in anesthetic practice for their sedative and analgesic effects. Tizanidine is a centrally acting a2-agonist with muscle relaxant, sedative and anxiolytic properties. This drug is widely used for the treatment of spasticity and has recently been used to treat musculoskeletal pain conditions.

Ultrasound (US) guidance during regional anesthesia practices has been a revolutionary advancement to improve success and safety of regional anesthesia. Analgesic effect of US guidance superficial cervical plexus block (SCPB) in patients undergoing thyroid surgery has not been reported yet.

The aim of this study was to evaluate the analgesic effect of preemptive oral single dose tizanidine and US guidance SCPB in patients undergoing elective thyroid surgery. The investigators hypothesis that: Tizanidine and US guided SCPB can reduce the pain scores, analgesic consumption, analgesic related side effects.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist's physiologic state I-III patients undergoing thyroidectomy

Exclusion Criteria:

* chronic pain
* bleeding disorders
* renal or hepatic insufficiency
* patients on chronic non-steroidal anti-inflammatory medications
* recurrent goiter
* emergency cases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Visual analog pain score | postoperative first hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at first hour postoperatively.
Visual analog pain score | postoperative second hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at second hour postoperatively.
Visual analog pain score | postoperative 4th hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at 4th hour postoperatively.
Visual analog pain score | postoperative 8th hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at 8th hour postoperatively.
Visual analog pain score | postoperative 12th hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS)score of 0-10 (0= no pain and 10= worst imaginable pain) at 12th hour postoperatively.
Visual analog pain score | postoperative 24th hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS)score of 0-10 (0= no pain and 10= worst imaginable pain) at 24th hour postoperatively.

SECONDARY OUTCOMES:
Opioid consumption | First 24 hours total opioid consumption

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ahiskalioglu, Ass.Prof., Principal Investigator — Ataturk University Anesthesiology and Reanimation
Locations (1):
- Ataturk University, Yakutiye, Erzurum, Turkey (Türkiye)

REFERENCES:
- [Background] Yazicioglu D, Caparlar C, Akkaya T, Mercan U, Kulacoglu H. Tizanidine for the management of acute postoperative pain after inguinal hernia repair: A placebo-controlled double-blind trial. Eur J Anaesthesiol. 2016 Mar;33(3):215-22. doi: 10.1097/EJA.0000000000000371. PMID 26555871
- [Background] Talakoub R, Abbasi S, Maghami E, Zavareh SM. The effect of oral tizanidine on postoperative pain relief after elective laparoscopic cholecystectomy. Adv Biomed Res. 2016 Feb 8;5:19. doi: 10.4103/2277-9175.175905. eCollection 2016. PMID 26962521
- [Background] Gurkan Y, Tas Z, Toker K, Solak M. Ultrasound guided bilateral cervical plexus block reduces postoperative opioid consumption following thyroid surgery. J Clin Monit Comput. 2015 Oct;29(5):579-84. doi: 10.1007/s10877-014-9635-x. Epub 2014 Oct 26. PMID 25344881
- [Derived] Ahiskalioglu A, Yayik AM, Oral Ahiskalioglu E, Dostbil A, Doymus O, Karadeniz E, Ari MA, Sengoz F, Alici HA, Celik EC. Ultrasound-guided bilateral superficial cervical block and preemptive single-dose oral tizanidine for post-thyroidectomy pain: a randomized-controlled double-blind study. J Anesth. 2018 Apr;32(2):219-226. doi: 10.1007/s00540-018-2468-x. Epub 2018 Feb 21. PMID 29468508